CLINICAL TRIAL: NCT00651170
Title: Can Ultrasound Predict Success of Median Nerve Block? Relationship Between Diffusion of Local Anesthetic and Effectiveness of a Nerve Block
Brief Title: Diffusion of Local Anesthetic After Median Nerve Block
Acronym: Echoalr
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/01
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Median Nerve
Keywords: Median block nerve; Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Median nerve block is widely practised, avoiding general anaesthesia in a number of cases and producing excellent post-operative analgesia in orthopedic surgery. Even realised by experienced anaesthetists,a failure rate of 5-15% is noticed. The principal aim of the study is to observe the local anesthetic solution diffusion after a conventional median nerve block technique using neurostimulation. The secondary objective is to compare diffusion and of block efficacy..

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective hand surgery requiring a median block nerve.

Exclusion Criteria:

* age lower than 18 years
* pregnancy
* contraindication to nerve block
* inability to read, write or speak French
* mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Anesthesic diffusion degree | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, Study Chair — Hopital Foch
Locations (2):
- France (2):
  - Hôpital Foch, Suresnes
  - Hôpital privé de l'Ouest Parisien, Trappes

IPD SHARING:
Plan to Share IPD: No